CLINICAL TRIAL: NCT03276572
Title: Phase I Dose-Escalation Trial of 225Ac-J591 in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Phase I Trial of 225Ac-J591 in Patients With mCRPC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Prostate Cancer Foundation (Other); United States Department of Defense (U.S. Federal Agency); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1706018281; 7R01CA207645-03 (NIH)
Record Dates: First submitted 2017-08-03; First posted 2017-09-08 (Actual); Results first posted 2022-12-06 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Subjects (Experimental): A single dose of 225Ac-J591 will be given to subjects with documented progressive metastatic CRPC.
  Interventions: Drug: 225Ac-J591

INTERVENTIONS:
Drug: 225Ac-J591 — 225Ac-J591 (13.3 KBq/Kg - 93.3 KBq/Kg or 0.36 uCi/Kg - 2.52 uCi/Kg) on day 1
  Other Names: 68Ga-PSMA-HBED-CC injection for PET/CT Scan on day 1 and at end of study

SUMMARY:
This is an open-label, single-center Phase I dose escalation study designed to determine the dose-limiting toxicity (DLT) and the maximum tolerated dose (MTD) of 225Ac-J591 in a single dose regimen.

DETAILED DESCRIPTION:
This clinical trial is for men with advanced prostate cancer. The purpose of this study is to find the highest dose level of the study drug, 225Ac-J591 that can be given without severe side effects. The research study is being done because the standard treatments for prostate cancer that has spread beyond the prostate gland are intended to minimize the adverse effects of the disease. These treatments, however, are not curative. Patients who choose to participate in this study will have a screening visit to determine whether or not they are eligible to participate in the study. The treatment phase is comprised of 8 visits over approximately 12 weeks. The study medication is called 225Ac-J591, and participants will receive an infusion of the study drug on the Treatment visit of the study. Upon completion of investigational treatment with single dose of 225Ac-J591, subjects will undergo 68Ga-PSMA-HBED-CC injection and same day PET/CT at the end of study visit to document treatment response. Subsequently survival data and additional treatment(s) information will be captured from their routine Standard of care (SOC) visits.During the other study visits, participants will undergo routine tests and procedures, such as physical examinations, and routine blood tests. Some blood tests will be done for research purposes only. After completion of therapy, participants may be contacted on a periodic basis to see how they are doing.

Key eligibility:

* Open to men age 18 and older.
* Diagnosis of progressive metastatic prostate cancer
* Have been previously treated for their disease with particular types of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of prostate
2. Documented progressive metastatic CRPC based on Prostate Cancer Working Group 3 (PCWG3) criteria, which includes at least one of the following criteria:

   1. PSA progression
   2. Objective radiographic progression in soft tissue
   3. New bone lesions
3. ECOG performance status of 0-2
4. Have serum testosterone < 50 ng/dL. Subjects must continue primary androgen deprivation with an LHRH analogue (agonist/antagonist) if they have not undergone bilateral orchiectomy.
5. Have previously been treated with at least one of the following:

   1. Androgen receptor signaling inhibitor (such as enzalutamide)
   2. CYP 17 inhibitor (such as abiraterone acetate)
6. Have previously received taxane chemotherapy, been determined to be ineligible for taxane chemotherapy by their physician, or refused taxane chemotherapy.
7. Age > 18 years
8. Patients must have normal organ and marrow function as defined below:

   1. Absolute neutrophil count >2,000 cells/mm3
   2. Hemoglobin ≥9 g/dL
   3. Platelet count >150,000 x 109/microliter
   4. Serum creatinine <1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 60 mL/min/1.73 m2 by Cockcroft-Gault
   5. Serum total bilirubin <1.5 x ULN (unless due to Gilbert's syndrome in which case direct bilirubin must be normal
   6. Serum AST and ALT <3 x ULN in absence of liver metastases; <5x ULN if due to liver metastases (in both circumstances, bilirubin must meet entry criteria)
9. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Implantation of investigational medical device ≤4 weeks of Cycle 1, Day 1 or current enrollment in oncologic investigational drug or device study
2. Use of investigational drugs ≤4 weeks or <5 half-lives of Cycle 1, Day 1 or current enrollment in investigational oncology drug or device study
3. Prior systemic beta-emitting bone-seeking radioisotopes
4. Known active brain metastases or leptomeningeal disease
5. History of deep vein thrombosis and/or pulmonary embolus within 1 month of C1D1
6. Other serious illness(es) involving the cardiac, respiratory, CNS, renal, hepatic or hematological organ systems which might preclude completion of this study or interfere with determination of causality of any adverse effects experienced in this study
7. Radiation therapy for treatment of PC ≤4 weeks of Day 1 Cycle 1
8. Patients on stable dose of bisphosphonates or Denosumab, which have been started no less than 4 weeks prior to treatment start, may continue on this medication, however patients are not allowed to initiate bisphosphonate/Denosumab therapy during the DLT-assessment period of the study.
9. Having partners of childbearing potential and not willing to use a method of birth control deemed acceptable by the principle investigator and chairperson during the study and for 1 month after last study drug administration
10. Currently active other malignancy other than non-melanoma skin cancer. Patients are considered not to have "currently active" malignancy if they have completed any necessary therapy and are considered by their physician to be at less than 30% risk of relapse.
11. Known history of known myelodysplastic syndrome

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult male patients of >18 years age with documented progressive metastatic CRPC
Enrollment: 32 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Tagawa, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Tulane Cancer Center Clinic, New Orleans, Louisiana
  - Weill Cornell Medical College, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tagawa ST, Thomas C, Sartor AO, Sun M, Stangl-Kremser J, Bissassar M, Vallabhajosula S, Huicochea Castellanos S, Nauseef JT, Sternberg CN, Molina A, Ballman K, Nanus DM, Osborne JR, Bander NH. Prostate-Specific Membrane Antigen-Targeting Alpha Emitter via Antibody Delivery for Metastatic Castration-Resistant Prostate Cancer: A Phase I Dose-Escalation Study of 225Ac-J591. J Clin Oncol. 2024 Mar 1;42(7):842-851. doi: 10.1200/JCO.23.00573. Epub 2023 Nov 3. PMID 37922438
- [Derived] Vlachostergios PJ, Niaz MJ, Skafida M, Mosallaie SA, Thomas C, Christos PJ, Osborne JR, Molina AM, Nanus DM, Bander NH, Tagawa ST. Imaging expression of prostate-specific membrane antigen and response to PSMA-targeted beta-emitting radionuclide therapies in metastatic castration-resistant prostate cancer. Prostate. 2021 Apr;81(5):279-285. doi: 10.1002/pros.24104. Epub 2021 Jan 19. PMID 33465252

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at at Weill Cornell Medicine New York Presbyterian and Tulane Medical Center.
Groups:
- 225Ac-J591 Cohort 1: Cohort 1: Participants were administered of 225Ac-J591 once at the dose level of 13.3 KBq/Kg - 0.36 Ci/Kg via intravenous infusion (IV). Participants were then followed until death for survival assessment
- 225Ac-J591 Cohort 2: Cohort 2: Participants were administered of 225Ac-J591 once at the dose level of 26.7 KBq/Kg - 0.72 Ci/Kg via intravenous infusion (IV). Participants were then followed until death for survival assessment.
- 225Ac-J591 Cohort 3: Cohort 3: Participants were administered of 225Ac-J591 once at the dose level of 40.0 KBq/Kg - 1.08 Ci/Kg via intravenous infusion (IV). Participants were then followed until death for survival assessment.
- 225Ac-J591 Cohort 4: Cohort 4: Participants were administered of 225Ac-J591 once at the dose level of 53.3 KBq/Kg - 1.44 Ci/Kg via intravenous infusion (IV). Participants were then followed until death for survival assessment.
- 225Ac-J591 Cohort 5: Cohort 5: Participants were administered of 225Ac-J591 once at the dose level of 66.7 KBq/Kg - 1.80 Ci/Kg via intravenous infusion (IV). Participants were then followed until death for survival assessment.
- 225Ac-J591 Cohort 6: Cohort 6: Participants were administered of 225Ac-J591 once at the dose level of 80.0 KBq/Kg - 2.16 Ci/Kg via intravenous infusion (IV). Participants were then followed until death for survival assessment.
- 225Ac-J591 Cohort 7: Cohort 7: Participants were administered of 225Ac-J591 once at the dose level of 93.3 KBq/Kg - 2.52 Ci/Kg via intravenous infusion (IV). Participants were then followed until death for survival assessment.
Period: Overall Study
Arm/Group | 225Ac-J591 Cohort 1 | 225Ac-J591 Cohort 2 | 225Ac-J591 Cohort 3 | 225Ac-J591 Cohort 4 | 225Ac-J591 Cohort 5 | 225Ac-J591 Cohort 6 | 225Ac-J591 Cohort 7
Started | 1 | 1 | 1 | 1 | 6 | 6 | 16
Completed | 1 | 1 | 1 | 1 | 6 | 5 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — In follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 225Ac-J591 Cohort 7: Cohort 7 with Expansion: Participants were administered of 225Ac-J591 once at the dose level of 93.3 KBq/Kg - 2.52 Ci/Kg via intravenous infusion (IV). Participants were then followed until death for survival assessment
- Total: Total of all reporting groups
Arm/Group | 225Ac-J591 Cohort 1 | 225Ac-J591 Cohort 2 | 225Ac-J591 Cohort 3 | 225Ac-J591 Cohort 4 | 225Ac-J591 Cohort 5 | 225Ac-J591 Cohort 6 | 225Ac-J591 Cohort 7 | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 6 | 6 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 1 | 2 | 5 | 8
  >=65 years | 1 | 1 | 1 | 1 | 5 | 4 | 11 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 1 | 1 | 1 | 1 | 6 | 6 | 16 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 1 | 1 | 6 | 6 | 16 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 1 | 1 | 1 | 1 | 5 | 6 | 15 | 30
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Dose Limiting Toxicities (DLT)
Description: Count of participants will be measured by the recommended phase II dose in utilizing the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 for DLTs.
Time Frame: Assessed from start of treatment to up to 8 weeks after first study drug administration.
Measure: Count of Participants; unit: Participants
Arm/Group | 225Ac-J591 Cohort 1 | 225Ac-J591 Cohort 2 | 225Ac-J591 Cohort 3 | 225Ac-J591 Cohort 4 | 225Ac-J591 Cohort 5 | 225Ac-J591 Cohort 6 | 225Ac-J591 Cohort 7
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0

2. Primary Outcome: Number of Subjects Who Reached Maximum Tolerated Dose (MTD)
Description: The MTD is the highest dose amongst the different dose-level cohorts in this study at which no more than 2 (33%) of the subjects in a cohort experience DLT.
Time Frame: Assessed from start of treatment to up to 8 weeks after first study drug administration.
Measure: Count of Participants; unit: Participants
Arm/Group | 225Ac-J591 Cohort 1 | 225Ac-J591 Cohort 2 | 225Ac-J591 Cohort 3 | 225Ac-J591 Cohort 4 | 225Ac-J591 Cohort 5 | 225Ac-J591 Cohort 6 | 225Ac-J591 Cohort 7
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 6 | 6 | 16
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Subjects With Prostate Specific Antigen (PSA) Response
Description: PSA will be analyzed through blood specimen collection
Time Frame: PSA was assessed at screening, and up to 6 months after first treatment with study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 225Ac-J591 Cohort 1 | 225Ac-J591 Cohort 2 | 225Ac-J591 Cohort 3 | 225Ac-J591 Cohort 4 | 225Ac-J591 Cohort 5 | 225Ac-J591 Cohort 6 | 225Ac-J591 Cohort 7
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 6 | 6 | 16
Participants | 0 | 1 | 1 | 0 | 3 | 3 | 10

4. Secondary Outcome: Number of Subjects With Circulating Tumor Cells (CTC) Response
Description: CTCs will be analyzed through blood specimen collection via CellSearch methodology lab testing
Time Frame: CTC was assessed at screening and 12 weeks after starting study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 225Ac-J591 Cohort 1 | 225Ac-J591 Cohort 2 | 225Ac-J591 Cohort 3 | 225Ac-J591 Cohort 4 | 225Ac-J591 Cohort 5 | 225Ac-J591 Cohort 6 | 225Ac-J591 Cohort 7
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 6 | 6 | 16
Participants | 1 | 1 | 1 | 1 | 5 | 5 | 8

5. Secondary Outcome: Number of Subjects With Radiographic (Imaging) Response
Description: Radiographic response rate by Response evaluation criteria in solid tumors (RECIST) criteria with Prostate Cancer Working Group 3 (PCWG3) modifications
Time Frame: Response were assessed for patients throughout their duration on the study, up to 3 years.
Measure: Count of Participants; unit: Participants
Arm/Group | 225Ac-J591 Cohort 1 | 225Ac-J591 Cohort 2 | 225Ac-J591 Cohort 3 | 225Ac-J591 Cohort 4 | 225Ac-J591 Cohort 5 | 225Ac-J591 Cohort 6 | 225Ac-J591 Cohort 7
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 6 | 6 | 16
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0

6. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From the start of treatment to progression, up to 3 years
Measure: Median (Full Range); unit: Days
Arm/Group | 225Ac-J591 Cohort 1 | 225Ac-J591 Cohort 2 | 225Ac-J591 Cohort 3 | 225Ac-J591 Cohort 4 | 225Ac-J591 Cohort 5 | 225Ac-J591 Cohort 6 | 225Ac-J591 Cohort 7
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 6 | 6 | 16
Days | 381 [381 to 381] | 56 [56 to 56] | 141 [141 to 141] | 60 [60 to 60] | 366 [95 to 940] | 242 [84 to 777] | 130 [54 to 334]

ADVERSE EVENTS:
Time Frame: Assessed throughout duration of participant on study, up to 3 years.
Arm/Group | 225Ac-J591 Cohort 1 | 225Ac-J591 Cohort 2 | 225Ac-J591 Cohort 3 | 225Ac-J591 Cohort 4 | 225Ac-J591 Cohort 5 | 225Ac-J591 Cohort 6 | 225Ac-J591 Cohort 7
All-Cause Mortality (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 1/1 | 6/6 | 6/6 | 15/16
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 3/6 | 2/6 | 8/16
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 1/1 | 6/6 | 6/6 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 225Ac-J591 Cohort 1 (N=1) | 225Ac-J591 Cohort 2 (N=1) | 225Ac-J591 Cohort 3 (N=1) | 225Ac-J591 Cohort 4 (N=1) | 225Ac-J591 Cohort 5 (N=6) | 225Ac-J591 Cohort 6 (N=6) | 225Ac-J591 Cohort 7 (N=16)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Any Pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin Increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 225Ac-J591 Cohort 1 (N=1) | 225Ac-J591 Cohort 2 (N=1) | 225Ac-J591 Cohort 3 (N=1) | 225Ac-J591 Cohort 4 (N=1) | 225Ac-J591 Cohort 5 (N=6) | 225Ac-J591 Cohort 6 (N=6) | 225Ac-J591 Cohort 7 (N=16)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 7 (7)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 5 (5) | 7 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 6 (6) | 12 (12)
Pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 4 (4) | 6 (6)
Xerostomia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 6 (6) | 5 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 6 (6) | 5 (5)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 6 (6) | 6 (6) | 15 (15)
Transaminase (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 6 (6) | 5 (5) | 8 (8)
Weight loss (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (4)
Dizziness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Dyspnea (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Generalized muscle soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased bilirubin (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT03276572/Prot_SAP_000.pdf